CLINICAL TRIAL: NCT06864962
Title: Efficacy and Safety Comparison of Renal Sympathetic Denervation Combined With Aorticorenal Ganglion Ablation vs. Renal Sympathetic Denervation Alone for the Treatment of Hypertension: A Multicenter, Prospective, Proof-of-concept Cohort Trials.
Brief Title: Renal Sympathetic Denervation Combined With Aorticorenal Ganglion Ablation for Treatment of Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The hospital ethics review for this study is currently underway, and participant recruitment will commence once the approval is granted.
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Shanghai Hongdian Medical CO., LTD (Industry)
Responsible Party: Principal Investigator, Yuehui Yin, Director of the Department, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RENATA-HTN
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Aorticorenal Ganglion; Renal Sympathetic Denervation; Autonomic Regulation; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSD group (Active Comparator): High-frequency stimulation (HFS) guided radiofrequency ablation from accessible branches to the opening of the renal artery.
  Interventions: Procedure: Renal sympathetic denervation
- RSD+ARGA group (Experimental): High-frequency stimulation (HFS) guided radiofrequency ablation from accessible branches to the opening of the renal artery, as well as HFS-guided ARG ablation.
  Interventions: Procedure: Renal sympathetic denervation plus aorticorenal ganglion ablation

INTERVENTIONS:
Procedure: Renal sympathetic denervation — Under the guidance of the 3-dimensional navigation system, HFS was performed from the accessible branches to the proximal (the ostium of renal artery) segments of the bilateral renal arteries, and the target ablation sites were identified by HFS-induced SBP elevation >5mmHg, and radiofrequency ablations were performed with a power setting of 8 to 12 Watts and a duration of 90 seconds. The endpoint of RSD was defined as the elimination or bluntness of HFS-induced SBP elevation response (≤5mmHg). If this was not achieved, ablation was repeated until the desired response was attained.
  Arms: RSD group
Procedure: Renal sympathetic denervation plus aorticorenal ganglion ablation — Following RSD, HFS was performed in the the junction area of abdominal aorta and renal arteries to recognize ARG. Radiofrequency ablations were performed with a power setting of 12 to 20 Watts and a duration of 90 seconds. The endpoint of ablation was defined as the elimination or bluntness of HFS-induced SBP elevation response (≤5mmHg). If this was not achieved, ablation was repeated until the desired response was attained.
  Arms: RSD+ARGA group

SUMMARY:
The purpose of this prospective cohort proof-of-concept trial is to compare the efficacy and safety of renal sympathetic denervation (RSD) plus aorticorenal ganglion ablation versus RSD alone in the treatment of uncontrolled primary hypertension.

DETAILED DESCRIPTION:
Currently, renal sympathetic denervation (RSD) has become the "third pillar" of hypertension treatment, following lifestyle interventions and pharmacological therapy. However, it still faces challenges such as limited and unstable blood pressure-lowering effects. One of the key factors contributing to the poor efficacy of the procedure is inadequate renal sympathetic nerve ablation, which is influenced by the complex renal artery anatomy and nerve network distribution. From a neuroanatomical perspective, aorticorenal ganglion (ARG) is a crucial hub for sympathetic nerve projection to the kidneys. We hypothesize that on the basis of RSD, additional ablation of aorticorenal ganglion can enhance the BP-lowering effect in patients with uncontrolled primary hypertension. Therefore, we plan to design the first multicenter, prospective, cohort, proof-of-concept trial to compare the efficacy and safety of RSD plus ARG ablation (ARGA) versus RSD alone in the treatment of uncontrolled primary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects;
* 18≤age≤70 years old;
* Primary hypertension;
* 24-hour ASBP ≥130mmHg after standard anti-hypertensive drug therapy;
* Arteries meet the criteria of catheter manipulation;
* Patient understands the purpose of this study, and is willing to participate and sign the informed consent;
* Patient is compliant and willing to complete clinical follow-up.

Exclusion Criteria:

* Abdominal aorta and renal arteries are not eligibility for catheter manipulation: 1) Renal artery stenosis >50% or any renal artery aneurysms on either side 2) History of renal artery percutaneous transluminal angioplasty (PTA), including balloon angioplasty and stenting; 3) abdominal aortic dissection, ulceration, or stenosis.
* eGFR <45ml/min/1.73m2 (MDRD formula)
* Hospitalized within one year due to hypertensive crisis
* Participated other clinical trials including both drug and medical device studies within 3 months enrollment
* Female with pregnant or lactating, or having plans for pregnancy within 1 year
* Patient with sleep apnea who needs chronic oxygen-breathing or mechanical ventilation support (for example, tracheostomy)
* Patients previously or currently suffering from one of the following diseases: 1) Essential pulmonary arterial hypertension; 2) Type I diabetes; 3) Severe cardiac valvular stenosis; 4) History of myocardial infraction (MI), unstable angina, syncope or cerebrovascular accidents within half year; 5) History of primary aldosteronism, pheochromocytoma, aorta stenosis, hyperthyroidism or hyperparathyroidism; 6) Any disease conditions interfering the measurement of blood pressure (for instance, severe peripheral artery diseases, abdominal artery aneurysm, hemorrhagic disorders such as thrombocytopenia, hemophilia and severe anemia); 7) Plans to have surgery or cardiovascular interventions within following 6 months; 8) Alcohol abuse or unknown drug dependence history; 9) Neuroticisms such as depression or anxiety disorders; 10) Non-compliant patients unable to finish the research per physician's requests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The change of 24-hour ambulatory systolic blood pressure | From enrollment to the end of treatment at 3 months

SECONDARY OUTCOMES:
The change of day-time ambulatory systolic blood pressure | From enrollment to the end of treatment at 3 months
The change of night-time ambulatory systolic blood pressure | From enrollment to the end of treatment at 3 months
The change of office systolic blood pressure | From enrollment to the end of treatment at 3 months
The change of drug burden index | From enrollment to the end of treatment at 3 months
Time of blood pressure controlling in target range | From enrollment to the end of treatment at 3 months

OTHER OUTCOMES:
The primary adverse events | From enrollment to the end of treatment at 3 months
  The primary adverse events was defined as the composite outcomes including all-cause mortality, end-stage renal disease, embolic events with end-organ damage, arterial perforation/dissection requiring intervention, hypertensive crisis requring hospitalization, new-onset renal stenosis (>70%)
The score of SF-36 | From enrollment to the end of treatment at 3 months
  SF-36: The Short-From-36 Health Survey
The score of GSRS | From enrollment to the end of treatment at 3 months
  GSRS: gastrointestinal symptom rating scale
The score of sexual function scale | From enrollment to the end of treatment at 3 months
  International Index of Erectile Function for male; Femal Sexual Function Index for female.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehui Yin, Professor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Nanan

IPD SHARING:
Plan to Share IPD: No